CLINICAL TRIAL: NCT05409027
Title: A Study to Assess 11 Beta-hydroxysteroid Dehydrogenase Type 1 Inhibition in Adipose Tissue by SPI-62
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sparrow Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SPI-62-CL-1001
Record Dates: First submitted 2022-03-23; First posted 2022-06-07 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Type 2 Diabetes Mellitus in Obese; Obesity; Type2Diabetes
MeSH Terms: conditions — Obesity | interventions — Glucocorticoids; Anti-Inflammatory Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Each subject will receive between 1 to 15 mg SPI-62 QD PO for up to 14 days.
  Each subject will receive up to 12 mcg cortisone-d8 SC during each of one or more study visits.
  Interventions: Drug: SPI-62; Drug: Cortisone-d8

INTERVENTIONS:
Drug: SPI-62 — SPI-62 is supplied as 1 mg tablets for oral dosing.
  Other Names: HSD-1 inhibitor
Drug: Cortisone-d8 — Cortisone-d8 is supplied as a 1 mcg/mL solution for infusion
  Other Names: Glucocorticoid and anti-inflammatory agent

SUMMARY:
This will be an exploratory, open-label study of 11β-hydroxysteroid dehydrogenase type 1 (HSD-1) inhibition by SPI-62 in obese subjects with type 2 diabetes mellitus (T2DM)

DETAILED DESCRIPTION:
The main objective of the study is to characterize the relationship between SPI-62 plasma concentration and adipose tissue inhibition of HSD-1 in obese subjects with T2DM.Additional objectives of the study are to characterize the relationship between adipose SPI-62 concentration and HSD-1 inhibition, to characterize the relationship between SPI-62 plasma concentration and liver inhibition of HSD-1, and to monitor the safety and tolerability of SPI-62, in obese subjects with T2DM. This will be a Phase I, open-label study in male and non-menstruating female subjects. Potential subjects will be screened to assess their eligibility to enter the study within 28 days prior to the first dose administration. Subjects will receive SPI-62 daily for up to 14 days. Subjects will also receive cortisone-d8, a mass-labeled HSD-1 substrate, by infusion during one or two confined study visits during the period of SPI-62 administration. Subjects may also receive cortisone-d8 during one to four additional confined study visits after cessation of SPI-62. Subjects will receive a follow-up call approximately 30 days after the last dose of study drug (SPI-62 or cortisone-d8). Results of population pharmacokinetic-pharmacodynamic modeling of data from this trial combined with those of prior trials will be reported separately from the Clinical Study Report.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-menstruating female
* 18 to 65 years of age
* BMI 30.0 to 45.0 kg/m2
* Diagnosis of T2DM for at least 3 months prior to the first dose of study drug.

Exclusion Criteria:

* Uncontrolled T2DM with glycated hemoglobin ≥9.5%.
* Any other current or prior medical condition expected to interfere with the conduct of the trial or the evaluation of its results.
* Any clinically significant abnormal laboratory value which cannot be explained by a known and permitted clinical condition.
* Positive urine drug screen (except tetrahydrocannabinol) or positive alcohol breath test result.
* Participation in a clinical trial involving administration of an investigational drug (new chemical entity) in the past 30 days or 5 half-lives, whichever is longer, or 90 days for a biological, prior to the first dose of study drug.
* Use of, or intent to use, any medications/products (prescription or over-the-counter) or herbal supplements within 4 weeks prior to the first dose of study drug, except those specifically allowed in the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2024-02-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (Cmax) | Days 1 through 14
  Pharmacokinetics of SPI-62 and its major metabolite AS2570469 by assessment of Observed Maximum Plasma Concentration (Cmax)

SECONDARY OUTCOMES:
Pharmacokinetics (tmax) | Days 1 through 14
  Pharmacokinetics of SPI-62 and its major metabolite AS2570469 by assessment of Time to Cmax (tmax)
Pharmacokinetics (AUC0-t) | Days 1 through 14
  Pharmacokinetics of SPI-62 and its major metabolite AS2570469 by assessment of Area Under the Curve over the dosing interval
Cortisone-d8 concentrations | Days 1 through 14
  individual values
Urinary HSD-1 Ratio | Days -1 to 15
  Individual values of the urinary HSD-1 ratio defined as (tetrahydrocortisol + allotetrahydrocortisol) / tetrahydrocortisone

CONTACTS AND LOCATIONS:
Overall Officials: David Katz, PhD, Study Director — Sparrow Pharmaceuticals
Locations (1):
- ProSciento, Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: No